CLINICAL TRIAL: NCT05908396
Title: An Open-Label, Multicenter, Phase 1 Study of IGM-2644 in Participants With Relapsed and/or Refractory Multiple Myeloma
Brief Title: Evaluation of IGM-2644 in Adults With Relapsed and/or Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company Decision
Sponsor: IGM Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IGM-2644-001
Record Dates: First submitted 2023-05-26; First posted 2023-06-18 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2023-08

CONDITIONS: Multiple Myeloma
Keywords: Relapsed and/or Refractory; Relapsed/Refractory Multiple Myeloma; CD38; Anti-CD3; Immunotherapy; monoclonal antibodies; bispecific; T-cell engager
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IGM-2644 Dose Escalation (Experimental): Participants will receive IGM-2644 via intravenous (IV) infusion weekly.
  Interventions: Drug: IGM-2644
- IGM-2644 Dose Expansion (Experimental): Participants will receive IGM-2644 via IV infusion at a dose and schedule to be determined after reviewing all available response and safety data.
  Interventions: Drug: IGM-2644

INTERVENTIONS:
Drug: IGM-2644 — IGM-2644 is an engineered, bispecific IgM antibody directed against CD3 and CD38. IGM-2644 is designed to bind to CD38 to selectively target and kill myeloma cancer cells through both T-cell dependent cellular toxicity (TDCC) and complement dependent cytotoxicity (CDC) activities.

SUMMARY:
This is a first in human, phase 1, multicenter, open-label study to determine the safety and tolerability of IGM-2644 as a single agent in participants with relapsed and/or refractory MM, for whom standard therapy does not exist, has proven to be ineffective or intolerable, or is considered inappropriate. Dose escalation and dose expansion cohorts will be enrolled to evaluate safety, preliminary efficacy, and further define a RP2D. The total length of the study, from screening of the first participant to the end of the study, is expected to be approximately 60 months.

DETAILED DESCRIPTION:
Patients will be enrolled in two stages: a dose-escalation stage and a dose expansion stage. The escalation stage will investigate single agent IGM-2644 safety and tolerability in patients with relapsed and/or refractory multiple myeloma. The dose expansion cohort(s) will further evaluate safety, PK/PD, and preliminary efficacy of the recommended phase 2 dose (RP2D).

IGM-2644 will be administered intravenously (IV).

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years at time of consent
* ECOG performance status of 0 or 1
* Relapsed and/or refractory multiple myeloma after ≥ 3 prior lines; Must have failed treatment with an IMiD, PI, and anti-CD38 therapy
* Measurable disease per the IMWG response criteria
* Adequate marrow and organ function without transfusion or growth factor support within 7 days prior to screening
* Willing and able to undergo bone marrow aspirate and biopsy per protocol

Exclusion Criteria:

* Inability to comply with study and follow-up procedures
* History of clinically significant primary amyloidosis, plasma cell leukemia, Waldenstrom macroglobulinemia or myelodysplastic syndrome
* Received chemotherapy, biologics, or small molecule therapy within 21 days or 5 half-lives, whichever is shorter
* Use of any non-approved or investigational agent ≤ 4 weeks prior to the first dose of study drug.
* Received last prior anti-CD38 monoclonal antibody treatment within 28 days before first planned dose of the study drug
* Current Grade > 1 toxicity, with the exception of Grade 2 peripheral neuropathy, alopecia, or toxicities from prior anti-tumor therapy that are considered irreversible
* Large-field radiotherapy within 28 days prior to Day 1 (radiation to a single site as concurrent therapy is allowed)
* Prior autologous stem cell transplant within 180 days prior to Day 1
* Prior allogeneic stem cell transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-08-29 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-02-16 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of IGM-2644 in participants with multiple myeloma, including estimation of the maximum tolerated dose (MTD) or maximum administered dose (MAD) | From Dose 1 through 30 days after the last dose of study treatment, approximately 14 months (each cycle is 21 days)
  Incidence of treatment-emergent AEs, SAEs, and DLT per NCI CTCAE v5.0

SECONDARY OUTCOMES:
Area Under the Curve (AUC) of IGM-2644 | At predefined intervals from Dose 1 through 30 days after the last dose of study treatment, approximately 14 months (each cycle is 21 days)
  Area Under the Curve (AUC) of IGM-2644 as a single agent
Clearance (CL) of IGM-2644 | At predefined intervals from Dose 1 through 30 days after the last dose of study treatment, approximately 14 months (each cycle is 21 days)
  Clearance (CL) of IGM-2644
Maximum Plasma Concentration (Cmax) of IGM-2644 | At predefined intervals from Dose 1 through 30 days after the last dose of study treatment, approximately 14 months (each cycle is 21 days)
  Maximum Plasma Concentration (Cmax) of IGM-2644 as a single agent
Half Life (HL) of IGM-2644 | At predefined intervals from Dose 1 through 30 days after the last dose of study treatment, approximately 14 months (each cycle is 21 days)
  Half Life (HL) of IGM-2644 as a single agent
Anti-Drug Antibodies (ADA) Formation | At predefined intervals from Dose 1 through 30 days after the last dose of study treatment, approximately 14 months (each cycle is 21 days)
  To evaluate the immunogenicity of IGM-2644 as a single agent
Objective Response Rate (ORR) | At predefined intervals from Dose 1 until documented disease progression, total overall study duration approximately 60 months
  To assess preliminary efficacy of IGM-2644 as a single agent, defined as the percentage of participants who achieve a confirmed complete response (CR), very good partial response (VGPR), or partial response (PR) per the International Myeloma Working Group (IMWG)
Duration of Response (DoR) | At predefined intervals from Dose 1 until documented disease progression, total overall study duration approximately 60 months
  For participants who demonstrate a confirmed complete response (CR), very good partial response (VGPR), or partial response (PR), defined as the time from the first documented response to the first documented disease progression or death, whichever occurs first.
Progression Free Survival (PFS) | At predefined intervals from Dose 1 until documented disease progression, total overall study duration approximately 60 months
  PFS is defined as the time from first dose to the first documented disease progression per IMWG criteria by investigator or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Manley, MD, Study Director — IGM Biosciences
Locations (5):
- United States (5):
  - City of Hope, Duarte, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Tennessee Oncology (SCRI), Nashville, Tennessee
  - Fred Hutchinson Cancer Research Center, Seattle, Washington